CLINICAL TRIAL: NCT01473953
Title: Investigation on Safety, Tolerability and Pharmacokinetics of Liraglutide-depot in Healthy Subjects. A Randomised, Double-blind, Placebo-controlled Trial Investigating Subcutaneously Single Dose Escalation of a Sustained Release Formulation of Liraglutide Lysine in Healthy Male Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of Liraglutide-depot in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9223-3928; U1111-1123-0547 (Other: WHO)
Record Dates: First submitted 2011-11-02; First posted 2011-11-17 (Estimated); Results first posted 2013-09-04 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1a: Lira-depot 2.25 mg (Experimental)
  Interventions: Drug: liraglutide-depot
- Cohort 2a: Lira-depot 6.75 mg (Experimental)
  Interventions: Drug: liraglutide-depot
- Cohort 3a: Lira-depot 15 mg (Experimental)
  Interventions: Drug: liraglutide-depot
- Cohort 4a: Lira-depot 30 mg (Experimental)
  Interventions: Drug: liraglutide-depot
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide-depot — Subjects will be randomised to receive a single dose of liraglutide-depot, at increasing dose levels, injected s.c./subcutaneously (under the skin). Progression to next dose level (max. 8) will be based on safety evaluation.
  Arms: Cohort 1a: Lira-depot 2.25 mg; Cohort 2a: Lira-depot 6.75 mg; Cohort 3a: Lira-depot 15 mg; Cohort 4a: Lira-depot 30 mg
Drug: placebo — Subjects will be randomised to receive a single dose of liraglutide-depot placebo, at increasing dose levels, injected s.c./subcutaneously (under the skin).
  Arms: Placebo

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to investigate the safety, tolerability and pharmacokinetics (exposure in the body) of liraglutide-depot in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 20 and 35 kg/m^2 (both inclusive) with a body weight of at least 60 kg
* Apart from being obese (BMI above 30 kg/m^2) the subject has to be considered generally healthy

Exclusion Criteria:

* Medical history of, or presence of, cancer, diabetes or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrine, haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders
* Clinical or laboratory findings which suggest that the subject cannot be considered generally healthy
* Prescription medicine and non-prescription medicine with few exceptions
* Current and prior history of alcohol or drug abuse
* Current smoking of more than 5 cigarettes per day
* Mental incapacity, language barriers, or unwillingness to comply with the protocol

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Evansville, Indiana, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at one site in Evansville, Indiana, USA.
Pre-assignment Details: It was a Novo Nordisk business decision, and not a decision due to safety concerns, not to continue the development of liraglutide depot. Therefore cohorts with liraglutide pre-treatment were not initiated based on review of pharmacokinetic data, and hence no analysis was done. So no subjects were enrolled for the outcome measure 6.
Groups:
- Cohort 1a: Lira-depot 2.25 mg: In cohort 1a a single subcutaneous dose of 2.25 mg liraglutide-depot was administered.
- Cohort 2a: Lira-depot 6.75 mg: In cohort 2a a single subcutaneous dose of 6.75 mg liraglutide-depot was administered.
- Cohort 3a: Lira-depot 15 mg: In cohort 3a a single subcutaneous dose of 15 mg liraglutide-depot was administered.
- Cohort 4a: Lira-depot 30 mg: In cohort 4a a single subcutaneous dose of 30 mg liraglutide-depot was administered.
- Placebo: In the placebo group a corresponding volume of liraglutide-depot placebo was administered subcutaneous (s.c.).
Period: Overall Study
Arm/Group | Cohort 1a: Lira-depot 2.25 mg | Cohort 2a: Lira-depot 6.75 mg | Cohort 3a: Lira-depot 15 mg | Cohort 4a: Lira-depot 30 mg | Placebo
Started | 6 | 6 | 6 | 5 | 8
Completed | 5 | 6 | 6 | 5 | 8
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1a: Lira-depot 2.25 mg | Cohort 2a: Lira-depot 6.75 mg | Cohort 3a: Lira-depot 15 mg | Cohort 4a: Lira-depot 30 mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 8 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (11.4) | 30.0 (12.6) | 29.8 (7.7) | 39.0 (8.4) | 28.5 (7.9) | 32.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 5 | 8 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs: AEs from 1st exposure (exp) until follow-up (FU) or AEs with onset before 1st exp increasing in severity up to the FU. Mild AEs: no or transient symptoms, no interference (inf) with subject's daily activities. Moderate AEs: marked symptoms, moderate inf with subject's daily activities. Severe AEs: considerable inf with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in death/ a life-threatening experience/ in-subject hospitalization/prolongation of existing hospitalisation; or persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Day 0 and up to 21 days after treatment
Population: The safety analysis set includes all subjects who were exposed to at least one dose of trial product. Subjects in the safety analysis set contribute to the evaluation 'as treated'.
Measure: Number; unit: events
Arm/Group | Cohort 1a: Lira-depot 2.25 mg | Cohort 2a: Lira-depot 6.75 mg | Cohort 3a: Lira-depot 15 mg | Cohort 4a: Lira-depot 30 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 8
events
  Total adverse events (AEs) | 3 | 3 | 4 | 21 | 13
  Serious AE | 0 | 0 | 0 | 0 | 0
  Severe AE | 0 | 0 | 0 | 1 | 0
  Moderate AE | 0 | 0 | 0 | 9 | 1
  Mild AE | 3 | 3 | 4 | 11 | 12
  Fatal AE | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Maximum Plasma Concentration of Liraglutide After a Single Dose of Liraglutide-depot
Time Frame: Day 0 through day 21 at 1,3,6,12,18, 24, 36, 48, 72, 96, 120, 168, 336, 504 hours post dose
Population: Full analysis set consisted of all subjects who were randomised and exposed to randomised treatment. This evaluation was not done on placebo cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | Cohort 1a: Lira-depot 2.25 mg | Cohort 2a: Lira-depot 6.75 mg | Cohort 3a: Lira-depot 15 mg | Cohort 4a: Lira-depot 30 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 0
pmol/L | 690 (52) [lower limit 52] | 2141 (25) [lower limit 25] | 6977 (62) [lower limit 62] | 40041 (35) [lower limit 35] |

3. Secondary Outcome: Time to Maximum Plasma Concentration of Liraglutide After a Single Dose of Liraglutide-depot
Time Frame: Day 0 through day 21 at 1,3,6,12,18, 24, 36, 48, 72, 96, 120, 168, 336, 504 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Cohort 1a: Lira-depot 2.25 mg | Cohort 2a: Lira-depot 6.75 mg | Cohort 3a: Lira-depot 15 mg | Cohort 4a: Lira-depot 30 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 0
hours | 15.13 (92.28) [lower limit 92.28] | 8.09 (55.78) [lower limit 55.78] | 13.74 (22.13) [lower limit 22.13] | 10.46 (24.62) [lower limit 24.62] |

4. Secondary Outcome: Area Under the Plasma Concentration Curve in the Period From the Time of Liraglutide-depot Administration to Infinity
Time Frame: Day 0 through day 21 at 1,3,6,12,18, 24, 36, 48, 72, 96, 120, 168, 336, 504 hours post dose
Population: Full analysis set consisted of all subjects who were randomised and exposed to randomised treatment. 1 subject was not included for this evaluation in the cohort 1a arm due to insufficient data. This evaluation was not done on placebo cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol.h/L
Arm/Group | Cohort 1a: Lira-depot 2.25 mg | Cohort 2a: Lira-depot 6.75 mg | Cohort 3a: Lira-depot 15 mg | Cohort 4a: Lira-depot 30 mg | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 0
pmol.h/L | 43840 (24) [lower limit 24] | 116935 (20) [lower limit 20] | 360000 (46) [lower limit 46] | 1443038 (22) [lower limit 22] |

5. Secondary Outcome: Area Under the Liraglutide Plasma Concentration Curve in the First Week Following Liraglutide-depot Administration for Subjects Without Liraglutide 6 mg/ml Pre-treatment
Time Frame: 1,3,6,12,18, 24, 36, 48, 72, 96, 120, 168 hours post dose
Population: Full analysis set consisted of all subjects who were randomised and exposed to randomised treatment. 1 subject was not included for this evaluation in the cohort 1a arm due to insufficient data. Cohorts with liraglutide pre-treatment were not initiated based on review of pharmacokinetic data, and hence no analysis was done.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol.h/L
Arm/Group | Cohort 1a: Lira-depot 2.25 mg | Cohort 2a: Lira-depot 6.75 mg | Cohort 3a: Lira-depot 15 mg | Cohort 4a: Lira-depot 30 mg | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 0
pmol.h/L | 37298 (27) [lower limit 27] | 114101 (20) [lower limit 20] | 316642 (46) [lower limit 46] | 1363187 (21) [lower limit 21] |

6. Secondary Outcome: Area Under the Plasma Concentration Curve in the First Week Following Liraglutide-depot Administration for Subjects With Liraglutide 6 mg/ml Pre-treatment
Time Frame: 0 to 168 hours after dosing
Population: Full analysis set consisted of all subjects who were randomised and exposed to randomised treatment. Cohorts with liraglutide pre-treatment were not initiated based on review of pharmacokinetic data, and hence no analysis was done.
Arm/Group | Cohort 1a: Lira-depot 2.25 mg | Cohort 2a: Lira-depot 6.75 mg | Cohort 3a: Lira-depot 15 mg | Cohort 4a: Lira-depot 30 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Subjects With Antibodies (Positive) or Without Antibodies (Negative) Against Liraglutide Observed at Pre-dose and at Last Follow-up
Time Frame: Day 0 and Day 21
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1a: Lira-depot 2.25 mg | Cohort 2a: Lira-depot 6.75 mg | Cohort 3a: Lira-depot 15 mg | Cohort 4a: Lira-depot 30 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 8
participants
  Positive | 0 | 0 | 0 | 0 | 0
  Negative | 6 | 6 | 6 | 5 | 8

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a timeframe of 7 days + 14 days follow up (Day 0 and up to 21 days after treatment)
Description: The safety analysis set includes all subjects who were exposed to at least one dose of trial product. Subjects in the safety analysis set contribute to the evaluation 'as treated'.
Arm/Group | Cohort 1a: Lira-depot 2.25 mg | Cohort 2a: Lira-depot 6.75 mg | Cohort 3a: Lira-depot 15 mg | Cohort 4a: Lira-depot 30 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/5 | 0/8
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 3/6 | 5/5 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1a: Lira-depot 2.25 mg (N=6) | Cohort 2a: Lira-depot 6.75 mg (N=6) | Cohort 3a: Lira-depot 15 mg (N=6) | Cohort 4a: Lira-depot 30 mg (N=5) | Placebo (N=8)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 3 (4)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site vasculitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.